CLINICAL TRIAL: NCT01782131
Title: A Phase 3 Randomized Study of the Efficacy and Safety of Posaconazole Versus Voriconazole for the Treatment of Invasive Aspergillosis in Adults and Adolescents (Phase 3; Protocol No. MK-5592-069)
Brief Title: A Study of the Safety and Efficacy of Posaconazole Versus Voriconazole for the Treatment of Invasive Aspergillosis (MK-5592-069)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06200; 5592-069 (Other: Merck); 2011-003938-14 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Fungal Infections; Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Mycoses; Invasive Pulmonary Aspergillosis | interventions — posaconazole; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posaconazole (POS) (Experimental): Participants received 300 mg posaconazole (POS) intravenous (IV) twice per day (BID) on Day 1, and then received 300 mg POS IV plus placebo IV once per day (QD) starting on Day 2 until clinically stable when participants transitioned to oral POS tablets plus oral placebo tablets QD for up to 12 weeks of treatment. Most participants were expected to initiate treatment with IV therapy and transition to oral therapy as clinically indicated, with some participants initiating treatment with oral therapy, per clinical judgment.
  Interventions: Drug: Posaconazole; Drug: Placebo
- Voriconazole (Active Comparator): Participants received 6 mg/kg voriconazole (VOR) IV twice per day (BID) on Day 1, and then received 4 mg/kg VOR IV BID on Day 2 until clinically stable when participants transitioned to oral therapy with VOR capsules or VOR placebo capsules BID for up to 12 weeks of treatment. Most participants were expected to initiate treatment with IV therapy and transition to oral therapy as clinically indicated, with some participants initiating treatment with oral therapy, per clinical judgment.
  Interventions: Drug: Voriconazole; Drug: Placebo

INTERVENTIONS:
Drug: Posaconazole — POS IV: Day 1: 300 mg BID Day 2-84: 300 mg QD POS oral: Day 1: 300 mg BID Day 2-84: 300 mg QD
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: Posaconazole (POS)
Drug: Voriconazole — VOR IV: Day 1: 6 mg/kg per body weight administered BID Day 2-84: 4 mg/kg per body weight administered BID VOR oral: Day 1: 300 mg BID Day 2-84: 200 mg BID
  Other Names: VFEND®
  Arms: Voriconazole
Drug: Placebo — Matching placebo received for Posaconazole (IV and oral) or Voriconazole (oral)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of posaconazole (POS) versus voriconazole (VOR) in the treatment of adults and adolescents with invasive aspergillosis (IA). The primary hypothesis is that the all-cause mortality through Day 42 in the POS treatment group is non-inferior to that in the VOR treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Weight >40 kg (88 lb) and ≤150 kg (330 lb); if between 13 and 14 years of age must weigh >= 50 kg (110 lb)
* Must meet the criteria for proven, probable, or possible IA as per 2008 European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) disease definitions at the time of randomization. Proven IA will include those participants with the demonstration of fungal elements (by cytology, microscopy, or culture) in diseased tissue (sterile sampling). Probable IA includes participants with at least 1 host factor, clinical criteria, as well as mycological criteria including both direct and indirect methods. Possible IA includes participants with at least 1 host factor and clinical criteria but without mycological criteria. A modification to the 2008 EORTC/MSG criteria regarding risk factors has been made to allow for the inclusion of participants with any duration of neutropenia as an acceptable inclusion host factor.
* If with possible IA at time of randomization must be willing or be in process of an ongoing diagnostic work up which is anticipated to result in a mycological diagnosis of proven or probable IA postrandomization.
* Must have a central line (e.g., central venous catheter, peripherally-inserted central catheter, etc.) in place or planned to be in place prior to beginning IV study therapy. If without central catheter access, must be clinically stable and able to receive oral study therapy.
* Acute IA defined as duration of clinical syndrome of <30 days.
* Must be willing to adhere to dosing, study visit schedule, and mandatory procedures as outlined in the protocol. The participant must be willing to continue on study therapy for up to 12 weeks and remain in the study through the 1-month follow-up visit.
* The participant must have the ability to transition to oral study therapy during the course of the study.
* Female participants of child-bearing potential must be using a medically accepted method of birth control before beginning study-drug treatment and agree to continue its use for 30 days after stopping study medication
* Is not taking prohibited antifungal prophylaxis or treatment

Exclusion Criteria:

* Chronic (>1 month duration) IA, relapsed/recurrent IA, or refractory IA which has not responded to antifungal therapy.
* Has pulmonary sarcoidosis, aspergilloma, or allergic bronchopulmonary aspergillosis (ABPA).
* Known mixed invasive mold fungal infection including Zygomycetes, and/or a known invasive Aspergillus fungal infection in which either study drug may not be considered active.
* Receipt of any systemic (oral, intravenous, or inhaled) antifungal therapy for this infection episode for 4 or more consecutive days (>= 96 hours) immediately before randomization.
* Developed the current episode of IA infection during receipt of >13 days of antifungal prophylaxis with an agent considered to be a mold-active antifungal agent.
* Receipt of posaconazole or voriconazole as empirical treatment for this infection for 4 days (96 hours) or more within the 15 days immediately before randomization.
* Has condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Known hypersensitivity or other serious adverse reaction to any azole antifungal therapy or to any other ingredient of the study medication used.
* Females who are pregnant, intend to become pregnant, or are nursing at the time of randomization.
* Known history of Torsade de Pointes, unstable cardiac arrhythmia or proarrhythmic conditions, or a history of recent myocardial infarction within 90 days of study entry.
* Has significant liver dysfunction
* Hepatic cirrhosis or a Child-Pugh score of C (severe hepatic impairment) at the time of randomization.
* Severe renal insufficiency (estimated creatinine clearance <20 mL/min) or on hemodialysis at the time of randomization or likely to require dialysis during the study.
* Known hereditary problem of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Acute symptomatic pancreatitis within 6 months of study entry or a diagnosis of chronic pancreatitis at the time of randomization.
* Active skin lesion consistent with squamous cell carcinoma at the time of randomization, or a current or prior history of malignant melanoma within 5 years of study entry.
* On artificial ventilation or receiving acute Continuous Positive Airway Pressure (CPAP)/Bilevel Positive Airway Pressure (BPAP) at the time of randomization.
* Known or suspected Gilbert's disease at the time of randomization.
* Requires treatment with other medications that cannot be stopped and for which there is a known contraindication to co-administration of one or more of the study drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Maertens JA, Rahav G, Lee DG, Haider S, Ramirez-Sanchez IC, Klimko N, Ponce-de-Leon A, Han S, Wrishko R, Winchell GA, Grandhi A, Waskin H; study investigators. Pharmacokinetic and Exposure Response Analysis of the Double-Blind Randomized Study of Posaconazole and Voriconazole for Treatment of Invasive Aspergillosis. Clin Drug Investig. 2023 Sep;43(9):681-690. doi: 10.1007/s40261-023-01282-7. Epub 2023 Sep 7. PMID 37676612
- [Derived] Maertens JA, Rahav G, Lee DG, Ponce-de-Leon A, Ramirez Sanchez IC, Klimko N, Sonet A, Haider S, Diego Velez J, Raad I, Koh LP, Karthaus M, Zhou J, Ben-Ami R, Motyl MR, Han S, Grandhi A, Waskin H; study investigators. Posaconazole versus voriconazole for primary treatment of invasive aspergillosis: a phase 3, randomised, controlled, non-inferiority trial. Lancet. 2021 Feb 6;397(10273):499-509. doi: 10.1016/S0140-6736(21)00219-1. PMID 33549194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After a screening phase of up to 7 days, 585 participants were enrolled/randomized, but only 575 began treatment (288 in the posaconazole [POS] group and 287 in the voriconazole [VOR] group).
Groups:
- Posaconazole: Participants received 300 mg posaconazole (POS) intravenous (IV) twice per day (BID) on Day 1, and then received 300 mg POS IV plus placebo IV once per day (QD) starting on Day 2 until clinically stable when participants transitioned to oral POS tablets plus oral placebo tablets QD for up to 12 weeks of treatment. Most participants were expected to initiate treatment with IV therapy and transition to oral therapy as clinically indicated, with some participants initiating treatment with oral therapy, per clinical judgment.
Period: Overall Study
Arm/Group | Posaconazole | Voriconazole
Started | 293 | 292
Treated | 288 | 287
Completed | 184 | 177
Not Completed | 109 | 115
Not completed — Death | 93 | 96
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Randomized but not treated | 5 | 5
Not completed — Reason not provided | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population included all participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole | Voriconazole | Total
Number analyzed (Participants) | 288 | 287 | 575
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (16.7) | 53.0 (15.9) | 53.3 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 231
  Male | 172 | 172 | 344
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 57 | 105
  Not Hispanic or Latino | 220 | 219 | 439
  Unknown or Not Reported | 20 | 11 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 6 | 10
  Asian | 62 | 60 | 122
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 194 | 192 | 386
  More than one race | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died Through Day 42 in the Intention to Treat Population
Description: The percentage of participants who died with posaconazole (POS) compared to voriconazole (VOR) in the first line treatment of invasive aspergillosis (IA) in the Intention to Treat (ITT) population through Day 42 was assessed.
Time Frame: Up to ~42 days
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 15.3 | 20.6
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Non-Inferiority — Based on Miettinen and Nurminen's method stratified by the risk for mortality/poor outcome (high risk, not high risk) and using Cochran-Mantel-Haenszel weighting scheme. The p-Value is based on the one-sided non-inferiority test. Non-inferiority of posaconazole vs. voriconazole is established if the upper limit of the 95% confidence interval is less than 10%; p < .0001, Miettinen and Nurminen; Estimated Difference in Percent = -5.3, 95% CI 2-sided [-11.6 to 1.0]

2. Secondary Outcome: Percentage of Participants Who Died Through Day 42 in the Full Analysis Set Population
Description: The percentage of participants who died with POS compared to VOR in the first line treatment of invasive aspergillosis (IA) in the Full Analysis Set (FAS) population through Day 42 was assessed.
Time Frame: Up to ~42 days
Population: The analysis population consisted of all randomized participants who have been classified as having proven or probable IA (based upon independent adjudication assessment using the modified 2008 European Organization for Research and Treatment of Cancer/Mycoses study group [EORTC/MSG] definitions) and received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Percentage of Participants | 19.0 | 18.7
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen and Nurminen's method stratified by the risk for mortality/poor outcome (high risk, not high risk) and using Cochran-Mantel-Haenszel weighting scheme; Estimated Difference in Percent = 0.3, 95% CI 2-sided [-8.2 to 8.8]

3. Secondary Outcome: Percentage of Participants Who Died Through Day 84 in the ITT Population
Description: The percentage of participants who died with POS compared to VOR in the first line treatment of invasive aspergillosis (IA) in the ITT population through Day 84 was assessed.
Time Frame: Up to ~84 days
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 28.1 | 30.7
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated Difference in Percent = -2.5, 95% CI 2-sided [-9.9 to 4.9]

4. Secondary Outcome: Percentage of Participants Who Died Through Day 84 in the FAS Population
Description: The percentage of participants who died with POS compared to VOR in the first line treatment of invasive aspergillosis (IA) in the FAS population through Day 84 was assessed.
Time Frame: Up to ~ 84 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Percentage of Participants | 34.4 | 31.0
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated Difference in Percent = 3.1, 95% CI 2-sided [-6.9 to 13.1]

5. Secondary Outcome: Percentage of Participants Achieving Global Clinical Response at Week 12 in the FAS Population
Description: The global clinical response of POS compared to VOR in the first line treatment of invasive aspergillosis (IA) was assessed. The percentage of participants achieving adjudicated global clinical response (complete or partial) at Week 12 was reported. Complete response was classified as survival with resolution of fungal disease evidence; Partial response was survival and improvement of fungal disease.
Time Frame: Up to 12 weeks (± 4 weeks)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Percentage of Participants | 42.3 | 46.2
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated Difference in Percent = -3.4, 95% CI 2-sided [-13.9 to 7.1]

6. Secondary Outcome: Percentage of Participants Achieving Global Clinical Response at Week 6 in the FAS Population
Description: The global clinical response of POS compared to VOR in the first line treatment of invasive aspergillosis (IA) was assessed. The percentage of participants achieving adjudicated global clinical response (complete or partial) at Week 6 was reported. Complete response was classified as survival with resolution of fungal disease evidence; Partial response was survival and improvement of fungal disease.
Time Frame: Up to 6 weeks (± 2 weeks)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Percentage of Participants | 44.8 | 45.6
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — [test comment as in outcome 2, analysis 1]; Difference in Percent = -0.6, 95% CI 2-sided [-11.2 to 10.1]

7. Secondary Outcome: Number of Participants Experiencing Mortality at Day 42, Day 84, and Day 114 in the FAS Population (Kaplan-Meier Time To Death Estimate)
Description: The number of participants experiencing mortality at Day 42, Day 84 and Day 114 in participants with proven or probable IA receiving POS versus VOR were assessed. The Kaplan-Meier estimate reports the number of participants who experienced death (all causes) through Day 114 or ~16 weeks. Participants who did not have any endpoint event until last visit or who were lost to follow-up and had no event were censored at the time of last available information (last study visit). For Day 42 and Day 84, missing or 'unable to determine' responses were considered as failures (dead).
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Participants
  Day 42 (missing responses were included as dead) | 31 | 32
  Day 84 (missing responses were included as dead) | 56 | 53
  Day 114 | 64 | 56
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Analysis of Time to All-Cause Mortality Through Day 114: Posaconazole vs. Voriconazole; Test type: Other; p = 0.2767, Kaplan-Meier — Based on Stratified Log-Rank method stratified by the risk for mortality/poor outcome (high risk, not high risk); From product-limit (Kaplan-Meier) method for censored data; Survival Rate in Percent = 60.7, 95% CI 2-sided [52.8 to 67.8]

8. Secondary Outcome: Number of Participants Who Died Due to Invasive Aspergillosis Through Day 42 in the FAS Population
Description: The number of participants who died due to IA receiving POS versus VOR through Day 42 was assessed.
Time Frame: Up to 42 days
Population: All randomized participants who died by Day 42 and who have been classified as having proven or probable IA (based upon independent adjudication assessment using the modified 2008 European Organization for Research and Treatment of Cancer/Mycoses study group [EORTC/MSG] definitions), and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Participants | 16 | 10
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen and Nurminen's method; Difference in Percent = 20.4, 95% CI 2-sided [-4.1 to 42.7]

9. Secondary Outcome: Number of Participants Who Died Due to Invasive Aspergillosis Through Day 84 in the FAS Population
Description: The number of participants who died due to IA receiving POS versus VOR in the FAS population through Day 84 was assessed.
Time Frame: Up to 84 days
Population: All randomized participants who died by Day 84 and who have been classified as having proven or probable IA (based upon independent adjudication assessment using the modified 2008 European Organization for Research and Treatment of Cancer/Mycoses study group [EORTC/MSG] definitions), and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 163 | 171
Participants | 22 | 14
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen and Nurminen's method; Difference in Percent = 11.3, 95% CI 2-sided [-6.9 to 28.6]

10. Secondary Outcome: Percentage of Participants With Tier 1 Treatment Emergent Adverse Events
Description: The percentage of participants with Tier 1 treatment-emergent adverse events (TEAEs) was determined. The Tier 1 TEAEs included hepatic safety (elevated aspartate serum transaminase [AST] or alanine serum transaminase [ALT] value ≥3x upper limit of normal (ULN) and an elevated total bilirubin value ≥2x ULN and, at the same time, an alkaline phosphatase value <2 ULN); central nervous system (CNS) and visual disturbances (eye disorders, nervous system disorders, psychiatric disorders), dermatologic reactions, and adrenal insufficiency or temporally associated TEAEs of hypotension.
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants
  Abnormal Hepatic Laboratory Value | 3.8 | 3.5
  CNS and Visual Disturbances | 32.3 | 35.9
  Dermatologic Reactions | 16.3 | 19.2
  Adrenal Insufficiency or Temporal Hypotension | 8.0 | 7.0
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Abnormal Hepatic Laboratory Value; Test type: Other; p = 0.8305, Miettinen & Nurminen; Difference in Percent = 0.3, 95% CI 2-sided [-2.9 to 3.6]
Statistical Analysis 2: Comparison: Posaconazole vs Voriconazole; CNS and Visual Disturbances; Test type: Other; p = 0.3633, Miettinen & Nurminen; Difference in Percent = -3.6, 95% CI 2-sided [-11.3 to 4.2]
Statistical Analysis 3: Comparison: Posaconazole vs Voriconazole; Dermatologic Reactions; Test type: Other; p = 0.3724, Miettinen & Nurminen; Difference in Percent = -2.8, 95% CI 2-sided [-9.1 to 3.4]
Statistical Analysis 4: Comparison: Posaconazole vs Voriconazole; Adrenal Insufficiency or Temporal Hypotension; Test type: Other; p = 0.6431, Miettinen & Nurminen; Difference in Percent = 1.0, 95% CI 2-sided [-3.4 to 5.5]

11. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product.
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 97.6 | 97.6
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-2.8 to 2.8]

12. Secondary Outcome: Percentage of Participants With at Least One Drug Related Adverse Event
Description: as for outcome 11
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 29.9 | 40.1
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen & Nurminen method; Difference in Percent = -10.2, 95% CI 2-sided [-17.9 to -2.4]

13. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event
Description: A serious adverse event (SAE) was an AE that resulted in death, was life threatening, required or prolonged an existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 61.8 | 59.9
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen & Nurminen method; Difference in Percent = 1.9, 95% CI 2-sided [-6.1 to 9.8]

14. Secondary Outcome: Percentage of Participants With at Least One Serious Drug Related Adverse Event
Description: An SAE was an AE that resulted in death, was life threatening, required or prolonged an existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to ~16 weeks (± 2 weeks)
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 5.6 | 7.0
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen & Nurminen method; Difference in Percent = -1.4, 95% CI 2-sided [-5.6 to 2.7]

15. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product.
Time Frame: Up to ~12 weeks
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole | Voriconazole
Number analyzed (Participants) | 288 | 287
Percentage of Participants | 32.3 | 35.5
Statistical Analysis 1: Comparison: Posaconazole vs Voriconazole; Test type: Other — Based on Miettinen & Nurminen method; Difference in Percent = -3.2, 95% CI 2-sided [-11.0 to 4.5]

16. Secondary Outcome: Steady State Average Concentration (Cavg) of Posaconazole With Food Intake
Description: The characterization of the pharmacokinetics (PK) parameters of POS was determined from plasma samples taken at steady-state after receiving oral tablet of POS. Steady-state Cavg, where Cavg is defined as area under the concentration time-curve from 0 to 24 hours (AUC0-24hr) divided by the dosing interval. Data is presented in POS group column only. No evaluation of food intake on the VOR capsule was presented.
Time Frame: Baseline, and at pre-dose on Day 7, Week 2, Week 4, Week 6, and Week 12
Population: The analysis population consisted of all randomized participants in the POS group only who received at least one dose of study treatment. Per protocol, the VOR group was not included in the analysis population because the food intake evaluation was limited to the POS group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 288
ng/mL
  Week 1: number analyzed (Participants) | 58
  Week 1 | 1625 (902.9)
  Week 2: number analyzed (Participants) | 64
  Week 2 | 1992 (1190)
  Week 4: number analyzed (Participants) | 67
  Week 4 | 1994 (956.3)
  Week 6: number analyzed (Participants) | 65
  Week 6 | 2005 (1333)
  Week 12: number analyzed (Participants) | 49
  Week 12 | 2169 (1255)

ADVERSE EVENTS:
Time Frame: Up to ~Week 16 (± 2 weeks)
Description: The analysis population was defined as all randomized participants who received at least one dose of study treatment. The analysis population for the all-cause mortality included all randomized participants.
Arm/Group | Posaconazole | Voriconazole
All-Cause Mortality (participants affected / at risk) | 99/293 | 99/292
Serious Adverse Events (participants affected / at risk) | 178/288 | 172/287
Other Adverse Events (participants affected / at risk) | 232/288 | 225/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=288) | Voriconazole (N=287)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (32) | 21 (26)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Accessory cardiac pathway (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neutropenic colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 2 (2) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 3 (3)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (9) | 5 (5)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 (2) | 2 (2)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 5 (5) | 3 (3)
Bacterial pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 6 (6) | 6 (6)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis pharyngeal (Infections and infestations) | 0 (0) | 1 (1)
Cerebral aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Citrobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis viral (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Disseminated cytomegaloviral infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 3 (4) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2)
Febrile infection (Infections and infestations) | 2 (2) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Hepatosplenic candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Mucormycosis (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 23 (27) | 12 (12)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Relapsing fever (Infections and infestations) | 1 (1) | 0 (0)
Renal graft infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 10 (10) | 7 (7)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 16 (16) | 16 (16)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 12 (12)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Precursor T-lymphoblastic lymphoma/leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Primary mediastinal large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 5 (5)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 2 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 5 (5)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (8)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=288) | Voriconazole (N=287)
Anaemia (Blood and lymphatic system disorders) | 23 (41) | 29 (46)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (24) | 18 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (28) | 17 (23)
Tachycardia (Cardiac disorders) | 11 (14) | 18 (23)
Abdominal pain (Gastrointestinal disorders) | 27 (31) | 24 (24)
Constipation (Gastrointestinal disorders) | 32 (36) | 23 (26)
Diarrhoea (Gastrointestinal disorders) | 52 (66) | 50 (57)
Nausea (Gastrointestinal disorders) | 65 (83) | 50 (63)
Vomiting (Gastrointestinal disorders) | 52 (64) | 38 (57)
Chest pain (General disorders) | 18 (19) | 11 (11)
Chills (General disorders) | 15 (19) | 8 (8)
Fatigue (General disorders) | 19 (20) | 7 (8)
Oedema peripheral (General disorders) | 32 (35) | 24 (27)
Pyrexia (General disorders) | 75 (122) | 69 (127)
Cytomegalovirus infection (Infections and infestations) | 15 (17) | 14 (16)
Pneumonia (Infections and infestations) | 14 (14) | 15 (15)
Alanine aminotransferase increased (Investigations) | 39 (49) | 34 (46)
Aspartate aminotransferase increased (Investigations) | 36 (46) | 34 (41)
Blood alkaline phosphatase increased (Investigations) | 21 (23) | 28 (33)
Blood bilirubin increased (Investigations) | 24 (38) | 20 (24)
Blood lactate dehydrogenase increased (Investigations) | 13 (17) | 17 (20)
Gamma-glutamyltransferase increased (Investigations) | 13 (15) | 15 (21)
Platelet count decreased (Investigations) | 15 (21) | 11 (18)
Decreased appetite (Metabolism and nutrition disorders) | 25 (25) | 14 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 15 (25) | 13 (27)
Hypokalaemia (Metabolism and nutrition disorders) | 78 (133) | 49 (72)
Hypomagnesaemia (Metabolism and nutrition disorders) | 29 (48) | 18 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (19) | 19 (26)
Hypophosphataemia (Metabolism and nutrition disorders) | 22 (24) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (20) | 13 (15)
Dizziness (Nervous system disorders) | 21 (22) | 12 (12)
Headache (Nervous system disorders) | 34 (45) | 24 (29)
Confusional state (Psychiatric disorders) | 8 (9) | 16 (16)
Insomnia (Psychiatric disorders) | 18 (19) | 16 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 24 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 24 (28)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31 (34) | 17 (17)
Rash (Skin and subcutaneous tissue disorders) | 19 (22) | 22 (32)
Hypertension (Vascular disorders) | 28 (33) | 23 (25)
Hypotension (Vascular disorders) | 17 (20) | 19 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media) that report any results of the trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT01782131/Prot_SAP_000.pdf